CLINICAL TRIAL: NCT00881868
Title: A Multi-Center, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Clobetasol Propionate Spray Versus Vehicle for the Management of Moderate to Severe Plaque Psoriasis of the Scalp
Brief Title: Clobetasol Propionate Spray Versus Vehicle Spray for the Management of Moderate to Severe Plaque Psoriasis of the Scalp
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: US10118
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2012-09

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clobex Spray (Active Comparator)
  Interventions: Drug: clobetasol propionate spray 0.05%
- Vehicle spray (Placebo Comparator)
  Interventions: Drug: Vehicle spray

INTERVENTIONS:
Drug: clobetasol propionate spray 0.05% — Apply enough product to cover affected areas topically twice daily at least 8 hours apart
  Other Names: Clobex® Spray 0.05%
  Arms: Clobex Spray
Drug: Vehicle spray — Apply enough product to cover affected areas topically twice daily at least 8 hours apart
  Arms: Vehicle spray

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of clobetasol propionate spray versus vehicle spray for the management of moderate to severe plaque psoriasis of the scalp.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of moderate to severe plaque psoriasis of the scalp

Exclusion Criteria:

* Subjects who need systemic treatment for their body psoriasis
* Subjects who have surface area involvement too large (>20% Body Surface Area [BSA]) that would require more than 50 grams per week of study product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (4):
- United States (4):
  - Dermatology Research Associates, Los Angeles, California
  - Hudson Dermatology, Evansville, Indiana
  - Research Division of The Skin Specialty Group, New York, New York
  - Dermatology Associates, PLLC, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on April 20, 2009 and the last subject was enrolled on November 17, 2009.
  Types of location: Investigative sites were located at private physician offices.
Pre-assignment Details: Wash-out period to baseline: 14 days: chemical hair process, steroid medication and/or ultraviolet B (UVB) treatment, calcipotriene, other vitamin D analogs, Anthralin/tar, all other anti-psoriasis medications; 4 wks: psoralen & UVA (PUVA) treatment & treatments other than biologics with possible efficacy on psoriasis; 12 wks: biological therapies
Period: Overall Study
Arm/Group | Clobex Spray | Vehicle Spray
Started | 41 | 40
Completed | 33 | 38
Not Completed | 8 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 4 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clobex Spray | Vehicle Spray | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (15.41) | 41.3 (13.72) | 43.7 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants in Each Category of the Scalp Psoriasis Individual Sign Scores (Scaling, Erythema and Plaque Elevation) at Baseline and Week 4
Description: Number of participants in each category of the Scalp Psoriasis Individual Sign Scores (Scaling, Erythema and Plaque Elevation) at baseline and end of treatment (week 4 or week 2 if GSS is Clear). Individual Sign Scores are evaluated on a scale from 0 - 4 (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe and 4 = Very Severe) with 0 being best and 4 being worst.
Time Frame: baseline to week 4
Measure: Number; unit: participants
Arm/Group | Clobex Spray | Vehicle Spray
Number analyzed (Participants) | 41 | 40
participants
  Scaling Baseline None (0) | 0 | 0
  Scaling Week 4 None (0) | 24 | 3
  Scaling Baseline Mild (1) | 4 | 2
  Scaling Week 4 Mild (1) | 15 | 9
  Scaling Baseline Moderate (2) | 22 | 26
  Scaling Week 4 Moderate (2) | 1 | 21
  Scaling Baseline Severe (3) | 12 | 11
  Scaling Week 4 Severe (3) | 1 | 7
  Scaling Baseline Very Severe (4) | 3 | 1
  Scaling Week 4 Very Severe (4) | 0 | 0
  Erythema Baseline None (0) | 0 | 1
  Erythema Week 4 None (0) | 24 | 3
  Erythema Baseline Mild (1) | 3 | 4
  Erythema Week 4 Mild (1) | 14 | 11
  Erythema Baseline Moderate (2) | 30 | 26
  Erythema Week 4 Moderate (2) | 3 | 20
  Erythema Baseline Severe (3) | 8 | 9
  Erythema Week 4 Severe (3) | 0 | 6
  Erythema Baseline Very Severe (4) | 0 | 0
  Erythema Week 4 Very Severe (4) | 0 | 0
  Plaque Elevation Baseline None (0) | 0 | 0
  Plaque Elevation Week 4 None (0) | 26 | 7
  Plaque Elevation Baseline Mild (1) | 7 | 2
  Plaque Elevation Week 4 Mild (1) | 13 | 12
  Plaque Elevation Baseline Moderate (2) | 19 | 27
  Plaque Elevation Week 4 Moderate (2) | 1 | 19
  Plaque Elevation Baseline Severe (3) | 13 | 11
  Plaque Elevation Week 4 Severe (3) | 1 | 2
  Plaque Elevation Baseline Very Severe (4) | 2 | 0
  Plaque Elevation Week 4 Very Severe (4) | 0 | 0

2. Secondary Outcome: Number of Participants in Each Category of the Extent of Scalp Involvement Index at Baseline and Week 4
Description: Number of participants in each category of the Extent of Scalp Involvement Index at end of treatment (week 4 or week 2 if GSS was Clear). The Extent of Scalp Involvement Index is evaluated on a scale from 0 - 5 (0 = None, 2 = <20%, 2 = 20-39%, 3 = 40-59%, 4 = 60-79% and 5 = 80-100%) with 0 being best and 5 being worst.
Time Frame: baseline to week 4
Measure: Number; unit: participants
Arm/Group | Clobex Spray | Vehicle Spray
Number analyzed (Participants) | 41 | 40
participants
  Extent of Scalp Involvement Baseline None | 0 | 0
  Extent of Scalp Involvement Week 4 None | 21 | 1
  Extent of Scalp Involvement Baseline <20% | 16 | 12
  Extent of Scalp Involvement Week 4 <20% | 16 | 16
  Extent of Scalp Involvement Baseline 20-39% | 5 | 6
  Extent of Scalp Involvement Week 4 20-39% | 4 | 12
  Extent of Scalp Involvement Baseline 40-59% | 12 | 14
  Extent of Scalp Involvement Week 4 40-59% | 0 | 4
  Extent of Scalp Involvement Baseline 60-79% | 6 | 5
  Extent of Scalp Involvement Week 4 60-79% | 0 | 5
  Extent of Scalp Involvement Baseline 80-100% | 2 | 3
  Extent of Scalp Involvement Week 4 80-100% | 0 | 2

3. Secondary Outcome: Number of Participants in Each Category of Pruritus at Baseline and Week 4
Description: Number of participants in each category of Pruritus at end of treatment (week 4 or week 2 if GSS was Clear). Pruritus is evaluated on a scale from 0 - 3 (0 = None, 1 = Mild, 2 = Moderate and 3 = Severe) with 0 being best and 3 being worst.
Time Frame: baseline to week 4
Measure: Number; unit: participants
Arm/Group | Clobex Spray | Vehicle Spray
Number analyzed (Participants) | 41 | 40
participants
  Pruritus Baseline None (0) | 4 | 1
  Pruritus Week 4 None (0) | 28 | 8
  Pruritus Baseline Mild (1) | 5 | 10
  Pruritus Week 4 Mild (1) | 12 | 14
  Pruritus Baseline Moderate (2) | 29 | 24
  Pruritus Week 4 Moderate (2) | 1 | 14
  Pruritus Baseline Severe (3) | 3 | 5
  Pruritus Week 4 Severe (3) | 0 | 4

4. Primary Outcome: Number of Participants Who Were a Success or Failure Based on the Global Severity Score (GSS) of Scalp Psoriasis From Baseline to End of Treatment (Week 4 or Week 2 if Clear)
Description: Number of participants who were a success or failure based on the Global Severity Score (GSS) of Scalp Psoriasis from baseline to end of treatment (Week 4 or Week 2 if Clear). GSS is evaluated on a scale from 0 - 5 (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe, 5 = Very Severe) with 0 being best and 5 being worst. Success is defined as Clear or Almost Clear. (Note: 5 Clobex Spray subjects and 0 Vehicle Spray subjects were Clear at week 2 and their results were carried forward to week 4).
Time Frame: baseline to week 4
Population: ITT, LOCF
Measure: Number; unit: participants
Arm/Group | Clobex Spray | Vehicle Spray
Number analyzed (Participants) | 41 | 40
participants
  Success | 35 | 5
  Failure | 6 | 35

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), if applicable.
Arm/Group | Clobex Spray | Vehicle Spray
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.